CLINICAL TRIAL: NCT03368573
Title: Optimising Medication Management in Children and Young People With Attention Deficit Hyperactivity Disorder (ADHD) Using an Objective Measure of Attention, Impulsivity and Activity (QbTest): a Feasibility Study
Brief Title: QbTest Utility for Optimising Treatment in ADHD (QUOTA)
Acronym: QUOTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottinghamshire Healthcare NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB-PG-1215-20026
Record Dates: First submitted 2017-11-22; First posted 2017-12-11 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2017-12

CONDITIONS: ADHD
Keywords: ADHD; Cognitive Assessment; QbTest; Medication; Feasibility
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Participants in the experimental arm (QbTest) protocol will also undergo standard assessment as usual plus a QbTest. If a QbTest was not conducted within 12 weeks prior to starting medication (as part of the ADHD diagnostic assessment procedure) the young person will sit a QbTest at baseline (off medication). Once on medication they will sit another QbTest 2-4 weeks after commencing medication and again 8-10 weeks later (and no later than 12 weeks).
  Participants in the control arm will undergo standard treatment as usual for ADHD. This will involve the clinician reviewing the child's symptom improvement once on medication and altering the dose according to their clinical judgement which may be informed by rating scales (completed by the parent, teacher and/or young person) and interviews with the parent and young person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention): Participants in the control arm will undergo standard treatment as usual for ADHD. This will involve the clinician reviewing the child's symptom improvement once on medication and altering the dose according to their clinical judgement which may be informed by rating scales (completed by the parent, teacher and/or young person) and interviews with the parent and young person.
- Experimental Arm (Experimental): Participants in the experimental arm (QbTest) protocol will also undergo standard assessment as usual plus a QbTest. If a QbTest was not conducted within 12 weeks prior to starting medication (as part of the ADHD diagnostic assessment procedure) the young person will sit a QbTest at baseline (off medication). Once on medication they will sit another QbTest 2-4 weeks after commencing medication and again 8-10 weeks later (and no later than 12 weeks).
  Interventions: Device: QbTest

INTERVENTIONS:
Device: QbTest — QbTest is a computerised assessment which takes approximately 20mins. The test combines a continuous performance test alongside an infrared camera which measures the participant's movements. The infrared camera measures motor activity of the participant whilst they undertake the task. During the test, the participant is presented with continuously changing stimuli. Embedded within these stimuli is a given target. Participants have to respond by pressing a hand-held button only when the target appears. Attention is measured through omission errors and reaction time to response. Impulsivity is assessed through commission errors and anticipatory errors. Motor activity is measured through head movements during the task. The test is approved by the FDA (Ref: K133382) and CE marked.
  Arms: Experimental Arm

SUMMARY:
Attention Deficit/Hyperactivity Disorder (ADHD) is a condition that affects 3-5% of young people under 18-years-old.

Young people with ADHD have difficulties with attention, impulsivity and hyperactivity that make it harder for them to learn, form relationships and prepare for adulthood. Clinical guidelines state that young people taking medication for ADHD should be closely monitored and have their medication reviewed regularly to ensure they receive the correct dose to improve their symptoms. However, many young people aren't monitored as closely as guidelines recommend. This can lead to lack of improvement or worsening of symptoms meaning that children may not experience the benefits of medication as quickly as they should. At the moment, assessing whether or not medication is working relies on the opinions of teachers and parents, collected through questionnaires. The difficulties of this are: differences of opinion between people, lack of information provided by them, and not returning the questionnaires. A test performed on a computer (QbTest) provides doctors with a report of the young person's symptoms and can therefore show whether medication is working. This may help doctors reach accurate decisions about medication dose more quickly, reducing the need for questionnaires. The study team met with families and young people with ADHD and medical experts and developed a procedure for using QbTest to measure medication effects. The study team will measure how well this procedure works in the real world by asking a group of young people to complete the test when they first start taking medication and at their follow-up appointments. The study team will ask doctors and families/young people for their opinions on the procedure.

The study team shall share our findings with other researchers and with the public by attending local support groups and providing summaries of the study results. The findings will be used to prepare for a future study.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the feasibility and acceptability of the study design using a feasibility RCT.

The end-points to assess this objective are:

* Acceptability of randomisation. The number of patients who do not participate and state randomisation as the reason for non-participation. The study team shall also monitor drop-out rates immediately after randomisation and the number of errors in randomisation at each site.
* Acceptability of study design. The number of eligible patients at each site and the numbers who consent to take part/withdraw. Withdrawal rates will be recorded alongside time point in the trial to ascertain acceptability of the study duration.
* Acceptability of outcome measures. Completion rates for outcomes to determine most appropriate methods of data collection.
* Acceptability/feasibility of protocol. Record non-adherence of healthcare professionals to the protocol and explore reasons.
* Feasibility of future RCT. Estimate the hours per week needed to run the RCT and therefore the number of research assistants/fellows required and time commitment required by HCPs.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 6-17 years (at the time of consent).
* Participant is willing and able to give informed consent for participation in the study (if over 16-years).
* Parental consent for children and young people aged under 16-years-old.
* Referred to CAMHS or Community Pediatric services and diagnosed with ADHD.
* Clinician and family (parent/carer and young person/child) agreement to commence stimulant medication for ADHD symptoms.

Exclusion Criteria:

* Unable to give informed consent
* Severe learning difficulty
* Not started on stimulant medication (either not started on medication at all or started on a non-stimulant medication)
* Non-fluent English

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
SNAP-IV | Follow up 2 (8-10 weeks)
  SNAP-IV is a short questionnaire designed to assess ADHD symptoms, with established validity, reliability and use in clinical and research settings. Completed by Parents and Teachers.

SECONDARY OUTCOMES:
SDQ | Baseline (0 weeks), Follow up 2 (8-10 weeks)
  The SDQ is a short, well validated and well used clinical and research measure that assesses a range of behavioural and emotional issues in children and young people. Completed by parents and teachers.
CHU9D | Baseline (0 weeks), Follow up 1 (2-4 weeks), Follow up 2 (8-10 weeks)
  a short (5 minute) measure of quality of life. The CHU9D has been designed for use with children and young people and is very easy to complete
CGI (Clinical Global Impressions Scale) | Baseline (0 weeks), Follow up 2 (8-10 weeks)
  Clinicians will be asked to complete the CGI. The CGI takes no longer than 5 minutes to complete and measures symptom severity and improvement due to medication.
Health Economic Outcome | Follow up 2 (8-10 weeks)
  Measure of use of Health Services
Side Effects Questionnaire | Follow up 1 (2-4 weeks) and Follow up 2 (8-10 weeks)
  To measure medication side effects
Medication adherence | Follow up 1 (2-4 weeks) and Follow up 2 (8-10 weeks)
  To look adherence to medication
Qualitative Interviews | Follow up 2 (8-10 weeks)
  To look at the acceptability of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Nottinghamshire Healthcare NHS Foundation Trust, Nottingham, United Kingdom

REFERENCES:
- [Derived] Williams L, Hall CL, Brown S, Guo B, James M, Franceschini M, Clarke J, Selby K, Vijayan H, Kulkarni N, Brown N, Sayal K, Hollis C, Groom MJ. Optimising medication management in children and young people with ADHD using a computerised test (QbTest): a feasibility randomised controlled trial. Pilot Feasibility Stud. 2021 Mar 16;7(1):68. doi: 10.1186/s40814-021-00788-1. PMID 33726855
- [Derived] Hall CL, Brown S, James M, Martin JL, Brown N, Selby K, Clarke J, Williams L, Sayal K, Hollis C, Groom MJ. Consensus workshops on the development of an ADHD medication management protocol using QbTest: developing a clinical trial protocol with multidisciplinary stakeholders. BMC Med Res Methodol. 2019 Jun 18;19(1):126. doi: 10.1186/s12874-019-0772-2. PMID 31215440
- [Derived] Hall CL, James M, Brown S, Martin JL, Brown N, Selby K, Clarke J, Vijayan H, Guo B, Sayal K, Hollis C, Groom MJ. Protocol investigating the clinical utility of an objective measure of attention, impulsivity and activity (QbTest) for optimising medication management in children and young people with ADHD 'QbTest Utility for Optimising Treatment in ADHD' (QUOTA): a feasibility randomised controlled trial. BMJ Open. 2018 Feb 15;8(2):e021104. doi: 10.1136/bmjopen-2017-021104. PMID 29453304